CLINICAL TRIAL: NCT05274555
Title: Reliability and Validity of the Turkish Version of the Upper Limb Short Questionnaire in Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Dilan Savaş, Physiotherapist, M.Sc., Dokuz Eylul University
Other Study IDs: 2019/07-65
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Duchenne Muscular Dystrophy; Upper Extremity Problem
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — The Upper Limb Short Questionnaire was administered by the researcher in face-to-face sessions with the children and their caregivers.
  The lower extremity functions and ambulation levels of the children were evaluated by the researcher using the Vignos Scale.
  The Brooke Upper Extremity Functional Rating Scale and ABILHAND-Kids were used to evaluate children's upper extremity functions.

SUMMARY:
Purpose: This study aimed to evaluate the construct validity and reliability of the Turkish version of the Upper Limb Short Questionnaire (ULSQ) in Duchenne muscular dystrophy (DMD).

Materials and methods: A total of 41 children with DMD have participated in the study. Upper and lower extremities functional levels were assessed with Vignos Scale and Brooke Upper Extremity Functional Rating Scale, respectively. The construct validity of the questionnaire was determined using the correlation between the ULSQ and ABILHAND-Kids. The Cronbach alpha value was calculated to determine internal consistency. To determine test-retest reliability, 17 randomly selected children were evaluated seven days after the first evaluation, and the "Intraclass Correlation Coefficient (ICC)" value was calculated.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with DMD, being between the ages of 5-18, not having any additional neurological disorder, volunteering to participate in the research

Exclusion Criteria:

* patients diagnosed after 10 years of age, patients who had never taken corticosteroids, and patients aged 14 years or older but were still ambulatory

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was planned as a methodological research. A total of 41 children with DMD between the ages of 5-18 were included in the study.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Upper Limb Short Questionnaire | 2 years
  The Upper Limb Short Questionnaire consists of questions about UE function (5 items), pain (6 items), and stiffness (3 items). ULSQ can be used as an identifier of arm-hand limitations during the clinical investigation. The total score changes between 0 and 14. Lower scores present children have more problems in the upper extremities.
ABILHAND-Kids | 2 years
  That evaluates upper extremity function according to 18 different activities performed by children. The total score calculates by summing the grades that children get from each item and change between 0 and 36. Lower scores present lower ability while higher scores indicate higher ability of the hand/upper extremity in the ABILHAND-Kids.
The Vignos Scale | 2 years
  This scale classifies patients' walking abilities in 10 grades ranging from 1 to 10. At the first level, the patient can walk and climb the steps without assistance, but at the last level, patient is confined to bed.
The Brooke Upper Extremity Functional Rating Scale | 2 years
  It classifies upper extremity function with 6 different levels based on the children's upper extremity movements. Level 1 means patient can start the movement with the arms at the sides and fully joins the hands above the head, Level 6 is defined as unable to raise their hands to their mouths and cannot use their hands functionally.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)